CLINICAL TRIAL: NCT03306277
Title: Phase 3, Open-Label, Single-Arm, Single-Dose Gene Replacement Therapy Clinical Trial for Patients With Spinal Muscular Atrophy Type 1 With One or Two SMN2 Copies Delivering AVXS-101 by Intravenous Infusion
Brief Title: Gene Replacement Therapy Clinical Trial for Participants With Spinal Muscular Atrophy Type 1
Acronym: STR1VE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Gene Therapies (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVXS-101-CL-303; 2020-000095-38 (EudraCT Number); COAV101A12302 (Other: Novartis Pharmaceuticals)
Record Dates: First submitted 2017-10-02; First posted 2017-10-11 (Actual); Results first posted 2020-07-16 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: SMA - Spinal Muscular Atrophy; Gene Therapy
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Zolgensma

STUDY DESIGN:
Intervention Model Description: One-time intravenous administration of onasemnogene abeparvovec-xioi.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Onasemnogene Abeparvovec-xioi (Experimental): One-time Intravenous administration of onasemnogene abeparvovec-xioi at the therapeutic dose.
  Interventions: Biological: Onasemnogene Abeparvovec-xioi

INTERVENTIONS:
Biological: Onasemnogene Abeparvovec-xioi — Non-replicating recombinant adeno-associated virus serotype 9 (AAV9) containing the complimentary deoxyribonucleic acid (cDNA) of the human SMN gene under the control of the cytomegalovirus (CMV) enhancer/chicken-β-actin-hybrid promoter (CB). The AAV inverted terminal repeat (ITR) has been modified to promote intramolecular annealing of the transgene, thus forming a double-stranded transgene ready for transcription.
  Other Names: Zolgensma

SUMMARY:
Phase 3 pivotal US trial studying open-label intravenous administration of onasemnogene abeparvovec-xioi in spinal muscular atrophy (SMA) Type 1 participants.

DETAILED DESCRIPTION:
Phase 3, open-label, single-arm, single-dose, study of onasemnogene abeparvovec-xioi (gene replacement therapy) in participants with spinal muscular atrophy (SMA) Type 1 who meet enrollment criteria and are genetically defined by nonfunctional survival motor neuron 1 gene (SMN1) with 1 or 2 copies of survival motor neuron 2 gene (SMN2). Fifteen (15) participants < 6 months (< 180 days) of age at the time of gene replacement therapy (Day 1) will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Participants with SMA Type 1 as determined by the following features: a. Diagnosis of SMA based on gene mutation analysis with bi-allelic SMN1 mutations (deletion or point mutations) and 1 or 2 copies of SMN2 (inclusive of the known SMN2 gene modifier mutation (c.859G>C))2
* The first 3 participants enrolled must meet the criteria for the Intent-To-Treat Population
* Participants must be < 6 months (< 180 days) of age at the time of onasemnogene abeparvovec-xioi infusion
* Participants must have a swallowing evaluation test performed prior to administration of gene replacement therapy
* Up-to-date on childhood vaccinations. Seasonal vaccinations that include palivizumab prophylaxis (also known as Synagis) to prevent respiratory syncytial virus (RSV) infections are also recommended in accordance with American Academy of Pediatrics
* Parent(s)/legal guardian(s) willing and able to complete the informed consent process and comply with study procedures and visit schedule

Exclusion Criteria:

* Previous, planned or expected scoliosis repair surgery/procedure during the study assessment period
* Pulse oximetry < 96% saturation at screening while the participant is awake or asleep without any supplemental oxygen or respiratory support, or for altitudes > 1000 m, oxygen saturation < 92% awake or asleep without any supplemental oxygen or respiratory support Pulse oximetry saturation may decrease to < 96% after screening provided that the saturation does not decrease by ≥ 4 percentage points
* Tracheostomy or current use or requirement of non-invasive ventilatory support averaging ≥ 6 hours daily over the 7 days prior to the screening visit; or ≥ 6 hours/day on average during the screening period or requiring ventilatory support while awake over the 7 days prior to screening or at any point during the screening period prior to dosing
* Participants with signs of aspiration/inability to tolerate non-thickened- liquids based on a formal swallowing test performed as part of screening. Participants with a gastrostomy tube who pass the swallowing test will be allowed to enroll in the study
* Participants whose weight-for-age is below the third percentile based on World Health Organization (WHO) Child Growth Standards
* Active viral infection (includes human immunodeficiency virus [HIV] or positive serology for hepatitis B or C, or Zika virus)
* Serious non-respiratory tract illness requiring systemic treatment and/or hospitalization within 2 weeks prior to screening
* Upper or lower respiratory infection requiring medical attention, medical intervention, or increase in supportive care of any manner within 4 weeks prior to screening
* Severe non-pulmonary/respiratory tract infection within 4 weeks before administration of gene replacement therapy or concomitant illness that creates unnecessary risks for gene replacement therapy such as: a. Major renal or hepatic impairment b. Known seizure disorder c. Diabetes mellitus d. Idiopathic hypocalcuria e. Symptomatic cardiomyopathy
* Known allergy or hypersensitivity to prednisolone or other glucocorticosteroids or their excipients
* Concomitant use of any of the following: drugs for treatment of myopathy or neuropathy, agents used to treat diabetes mellitus, or ongoing immunosuppressive therapy, plasmapheresis, immunomodulators such as adalimumab, immunosuppressive therapy within 3 months prior to gene replacement therapy
* Anti-adeno-associated virus serotype 9 (AAV9) antibody titer > 1:50 as determined by Enzyme-linked Immunosorbent Assay (ELISA) binding immunoassay. Should a potential participant demonstrate Anti-AAV9 antibody titer > 1:50, he or she may receive retesting within 30 days of the screening period and will be eligible to participate if the Anti-AAV9 antibody titer upon retesting is ≤ 1:50
* Clinically significant abnormal laboratory values (gamma glutamyl- transpeptidase [GGT], ALT, and AST > 3 × ULN, bilirubin ≥ 3.0 mg/dL, creatinine ≥ 1.0 mg/dL, hemoglobin [Hgb] < 8 or > 18 g/dL; white blood cell [WBC] > 20,000 per cmm) prior to gene replacement therapy
* Participation in recent SMA treatment clinical study (with the exception of observational Cohort studies or non-interventional studies) or receipt of an investigational or commercial compound, product, or therapy administered with the intent to treat SMA at any time prior to screening for this study. Oral β-agonists must be discontinued at least 30 days before gene therapy dosing. Inhaled albuterol specifically prescribed for the purposes of respiratory (bronchodilator) management is acceptable and not a contraindication at any time prior to screening for this study
* Expectation of major surgical procedures during the study assessment period
* Parent(s)/legal guardian(s) unable or unwilling to comply with study procedures or inability to travel for repeat visits
* Parent(s)/legal guardian(s) unwilling to keep study results/observations confidential or to refrain from posting confidential study results/observations on social media sites
* Parent(s)/legal guardian(s) refuses to sign consent form
* Gestational age at birth < 35 weeks (245 days)

Max Age: 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Stanford University, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Hospital, Orlando, Florida
  - Ann and Robert H Lurie Children's Hospital, Chicago, Illinois
  - Johns Hopkins Pediatric Neurology, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington Unviersity School of Medicine, St Louis, Missouri
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Wisconsin (Madison), Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.
URL: https://www.clinicalstudydatarequest.com/.

REFERENCES:
- [Derived] Day JW, Mendell JR, Mercuri E, Finkel RS, Strauss KA, Kleyn A, Tauscher-Wisniewski S, Tukov FF, Reyna SP, Chand DH. Clinical Trial and Postmarketing Safety of Onasemnogene Abeparvovec Therapy. Drug Saf. 2021 Oct;44(10):1109-1119. doi: 10.1007/s40264-021-01107-6. Epub 2021 Aug 12. PMID 34383289
- [Derived] Day JW, Finkel RS, Chiriboga CA, Connolly AM, Crawford TO, Darras BT, Iannaccone ST, Kuntz NL, Pena LDM, Shieh PB, Smith EC, Kwon JM, Zaidman CM, Schultz M, Feltner DE, Tauscher-Wisniewski S, Ouyang H, Chand DH, Sproule DM, Macek TA, Mendell JR. Onasemnogene abeparvovec gene therapy for symptomatic infantile-onset spinal muscular atrophy in patients with two copies of SMN2 (STR1VE): an open-label, single-arm, multicentre, phase 3 trial. Lancet Neurol. 2021 Apr;20(4):284-293. doi: 10.1016/S1474-4422(21)00001-6. Epub 2021 Mar 17. PMID 33743238
- See also: sponsor company website — http://AveXis.com
- See also: Novartis Results Record — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17657
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1219

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22 participants were recruited across 16 study centers in the United States.
Pre-assignment Details: A screening period of up to 30 days occurred before treatment.
Period: Overall Study
Arm/Group | Onasemnogene Abeparvovec-xioi
Started | 22
Completed | 19
Not Completed | 3
Not completed — Death | 1
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Onasemnogene Abeparvovec-xioi
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 3.7 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 11
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 22
Patient reported hospitalizations [Number; unit: participants]
  Yes | 17
  No | 5
Weight at baseline [Mean (Standard Deviation); unit: kg] | 5.8 (1.1)
Height/length at baseline [Mean (Standard Deviation); unit: cm] | 61.3 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Achievement of Independent Sitting for at Least 30 Seconds
Description: Independent sitting is defined as sitting up straight with head erect for at least 30 seconds.
  This endpoint is a co-primary endpoint. The two co-primary efficacy endpoints were assessed in sequence: The endpoint of functional independent sitting was assessed first and, only when this assessment met statistical significance, was the endpoint of event-free survival assessed.
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Onasemnogene Abeparvovec-xioi
Number analyzed (Participants) | 22
Participants | 13
Statistical Analysis 1: Comparison: Onasemnogene Abeparvovec-xioi; This comparison is made to an assumed rate of zero 0 (or as low as 0.1%). By definition, children with spinal muscular atrophy Type 1 are never able to sit independently; Test type: Superiority; p < 0.0001, One-sided Exact Binomial Test

2. Primary Outcome: Event-free Survival
Description: Survival is defined by the avoidance of combined endpoint of either death or permanent ventilation, which is defined by tracheostomy or by the requirement of ≥ 16 hours of respiratory assistance per day for ≥ 14 consecutive days in the absence of an acute reversible illness, excluding perioperative ventilation. Permanent ventilation is considered a surrogate for death. An acute reversible illness is defined as any condition other than SMA that results in increased medical intervention.
  The endpoint is a co-primary endpoint. The two co-primary efficacy endpoints were assessed in sequence: The endpoint of functional independent sitting was assessed first and, only when this assessment met statistical significance was the survival endpoint assessed.
Time Frame: 14 months
Measure: Count of Participants; unit: Participants
Arm/Group | Onasemnogene Abeparvovec-xioi
Number analyzed (Participants) | 22
Participants | 20
Statistical Analysis 1: Comparison: Onasemnogene Abeparvovec-xioi; This comparison is made against the results from the age and gender-matched control participants selected from existing natural history data sets (PNCR) [Neurol. 2014; 83(9):810-817]; Test type: Superiority; p < 0.0001, Fisher Exact; Data for the current study were compared to historical control data (Finkel et al,2014 - PubMed 25080519) where event-free survival was 6 out of 23 participants (26.1%) at 14 months of age

3. Secondary Outcome: Ability to Thrive
Description: Ability to thrive is defined as achieving all of the following at 18 months of age:
  * does not receive nutrition through mechanical support or other non-oral method
  * ability to tolerate thin liquids as demonstrated through a formal swallowing test
  * maintains weight
  This is a co-secondary endpoint. The two co-secondary endpoints were assessed in sequence: The endpoint of ability to thrive was assessed first and, only when this assessment met statistical significance was the endpoint of ventilatory support independence assessed.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Onasemnogene Abeparvovec-xioi
Number analyzed (Participants) | 22
Participants | 9

4. Secondary Outcome: Ventilatory Support Independence
Description: Ventilatory support independence is defined as requiring no daily ventilator support/usage at 18 months of age, excluding acute reversible illness and perioperative ventilation, through assessment of actual usage data captured from the device (Phillips Trilogy BiPAP device). This endpoint is derived solely from the Phillips Trilogy BiPAP device.
  This is a co-secondary endpoint. The two co-secondary endpoints were assessed in sequence: The endpoint of ability to thrive was assessed first and, only when this assessment met statistical significance was the endpoint of ventilatory support independence assessed.
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Onasemnogene Abeparvovec-xioi
Number analyzed (Participants) | 22
Participants | 18

ADVERSE EVENTS:
Time Frame: Up to 18 months
Arm/Group | Onasemnogene Abeparvovec-xioi
All-Cause Mortality (participants affected / at risk) | 1/22
Serious Adverse Events (participants affected / at risk) | 10/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Onasemnogene Abeparvovec-xioi (N=22)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Human metapneumovirus test positive (Investigations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Cyanosis (Cardiac disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Device malfunction (Product Issues) | 1 (1)
Abnormal weight gain (Metabolism and nutrition disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Feeding disorder (Metabolism and nutrition disorders) | 1 (1)
Bronchiolitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 (2)
Bacterial tracheitis (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (2)
Sepsis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Onasemnogene Abeparvovec-xioi (N=22)
Diastolic hypertension (Vascular disorders) | 2 (2)
Pyrexia (General disorders) | 12 (26)
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Contusion (Injury, poisoning and procedural complications) | 4 (4)
Arthropod bite (Injury, poisoning and procedural complications) | 3 (7)
Aspartate aminotransferase increased (Investigations) | 6 (9)
Alanine aminotransferase increased (Investigations) | 5 (8)
Blood creatine phosphokinase MB increased (Investigations) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (2)
Weight decreased (Investigations) | 2 (2)
Pericardial effusion (Cardiac disorders) | 2 (2)
Pectus excavatum (Congenital, familial and genetic disorders) | 3 (3)
Asphyxiating thoracic dystrophy (Congenital, familial and genetic disorders) | 2 (2)
Cryptorchism (Congenital, familial and genetic disorders) | 2 (2)
High arched palate (Congenital, familial and genetic disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 6 (10)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory track congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Muscle contractions involuntary (Nervous system disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 9 (11)
Teething (Gastrointestinal disorders) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (8)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (3)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Scoliosis (Musculoskeletal and connective tissue disorders) | 9 (12)
Deformity thorax (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint contracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Kyphosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Torticollis (Musculoskeletal and connective tissue disorders) | 2 (2)
Feeding disorder (Metabolism and nutrition disorders) | 3 (4)
Weight gain poor (Metabolism and nutrition disorders) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 11 (28)
Conjunctivitis (Infections and infestations) | 3 (3)
Otitis media (Infections and infestations) | 3 (4)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 (3)
Gastroenteritis (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)

LIMITATIONS AND CAVEATS:
The complete results are available via this link: https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17657

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release and has right to request changes to communications regarding trial results for a period that is more or equal to 30 days but less than or equal to 150 days from the time submitted to the Sponsor for review in order to either delete references to Sponsor's Confidential Information or delay such results communications to permit Sponsor to obtain appropriate Intellectual Property protection as set forth in the agreement.

DOCUMENTS (2):
  • Study Protocol (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT03306277/Prot_001.pdf
  • Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT03306277/SAP_000.pdf